CLINICAL TRIAL: NCT05327322
Title: The Impact of Diet Quality and Calorie Restriction on Physical Function and Patient Reported Outcomes in Multiple Sclerosis
Brief Title: Functional Outcomes From Diets in Multiple Sclerosis
Acronym: FOOD_for_MS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Washington University School of Medicine (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Brooks C. Wingo, PhD, Associate Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 300009050; CDMRP-MS210011 (Other Grant/Funding Number: US Department of Defense)
Record Dates: First submitted 2022-03-24; First posted 2022-04-14 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-04

CONDITIONS: Relapsing Remitting Multiple Sclerosis; Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive | interventions — Glycemic Load; Caloric Restriction; Behavior Therapy

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to follow either a low GL or standard GL diet for 32 weeks. For the first 16 weeks, both groups will eat enough calories to maintain baseline weight. During the second 16 weeks, both groups will reduce calorie intake by 500 kcal/day,
Who Masked: Outcomes Assessor
Masking Description: All staff collecting outcomes data will be randomized to treatment group (low GL vs standard GL).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low Glycemic Load (Experimental): This group will be prescribed a daily GL of <45 points/1000 kcal and 25% of daily calorie intake from carbohydrates. This group will be provided few processed foods. During the first 16 weeks, this group will eat enough calories to maintain baseline weight, and will reduce daily calorie intake by 500 kcal/day in the second 16 weeks.
  Interventions: Behavioral: Glycemic load; Behavioral: Calorie restriction; Behavioral: Behavioral support
- Standard Glycemic Load (Active Comparator): This group will be prescribed a daily GL of >75 points/1000kcal and 60% of daily calorie intake from carbohydrates. This group will be provided more processed foods than the low GL group. During the first 16 weeks, this group will eat enough calories to maintain baseline weight, and will reduce daily calorie intake by 500 kcal/day in the second 16 weeks.
  Interventions: Behavioral: Glycemic load; Behavioral: Calorie restriction; Behavioral: Behavioral support

INTERVENTIONS:
Behavioral: Glycemic load — Participants will be provided food to meet GL prescription for the duration of the trial.
Behavioral: Calorie restriction — Participants will be provided food to meet their prescribed daily calorie intake for the duration of the trial (weight stable in first 16 weeks, weight loss in second 16 weeks).
Behavioral: Behavioral support — All participants will receive behavioral supports in the form of email, text, information pages and weekly calls from the study staff to maximize adherence.

SUMMARY:
The purpose of this study is to test the effects of two dietary interventions, glycemic load and calorie restriction, on physical function, cognition, pain, fatigue, mood, and anxiety in adults with multiple sclerosis (MS). The investigators will also explore the how the diet interventions impact inflammation, immunity, and metabolic biomarkers.

DETAILED DESCRIPTION:
100 participants will be randomized 1:1 to follow either a low glycemic load (GL) or standard GL diet for 32 weeks. For the first 16 weeks, all participants will eat enough calories to maintain their baseline weight. During the second 16 weeks, all participants will reduce calorie intake by 500kcal/day, with a goal of losing 5-10% of initial body weight. Participants will complete data collection at baseline (prior to randomization), at 17 weeks (after the weight stable phase) and again after completing the calorie restriction phase.

All participants will receive meal plans and groceries for the duration of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with RRMS or SPMS
* BMI 25-50 kg/m2 (overweight/obese)
* EDSS ≤6.5 (able to walk 100m with or without assistance)
* If on disease-modifying treatment (DMT), stable for 6 months
* If not on DMT, no DMT in previous 6 months
* No expected change to DMT in next 34 weeks
* Responsible for food preparation or have input into food preparation

Exclusion Criteria:

* MS relapse in previous 30 days
* Unable to walk 25 feet with or without assistive device
* Pregnant or breastfeeding
* Current use of insulin or sulfonylurea agents
* Score indicating low cognitive functioning on the Telephone Interview for Cognitive Status (TICS-m) assessment
* Actively engaged in a weight loss program or unwilling to follow assigned dietary pattern
* Unable to receive, store, or prepare food according to diet plan
* Medical contraindication to either treatment or control diet (including severe allergies that cannot be accommodated within either group)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-20 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Multiple Sclerosis Functional Composite (MSFC) | Baseline
  The MSFC includes a timed T25FW, 9-hole peg test (9HPT), and the Paced Auditory Serial Addition Test (PASAT).
Multiple Sclerosis Functional Composite (MSFC) | 17 weeks
  The MSFC includes a timed T25FW, 9-hole peg test (9HPT), and the Paced Auditory Serial Addition Test (PASAT).
Multiple Sclerosis Functional Composite (MSFC) | 34 weeks
  The MSFC includes a timed T25FW, 9-hole peg test (9HPT), and the Paced Auditory Serial Addition Test (PASAT).

SECONDARY OUTCOMES:
Brief International Cognitive Assessment for MS (BICAMS) | Baseline
  The BICAMS includes the Single Digit Modalities Test, California Verbal Learning Test, and Brief Visuospatial Memory Test
Brief International Cognitive Assessment for MS (BICAMS) | 17 weeks
  The BICAMS includes the Single Digit Modalities Test, California Verbal Learning Test, and Brief Visuospatial Memory Test
Brief International Cognitive Assessment for MS (BICAMS) | 34 weeks
  The BICAMS includes the Single Digit Modalities Test, California Verbal Learning Test, and Brief Visuospatial Memory Test
Patient reported outcomes: Hospital Anxiety and Depression Scale (HADS) | Baseline
  The HADS contains 14 items that measure the frequency of anxiety and depressive symptoms over the past week. The anxiety questions are scaled 0-3 with 0 representing higher anxiety to 3 representing no anxiety. The depression questions are scaled from 0 indicating no depression to 3 indicating more signs of depression.
Patient reported outcomes: Hospital Anxiety and Depression Scale (HADS) | 17 weeks
  The HADS contains 14 items that measure the frequency of anxiety and depressive symptoms over the past week. The anxiety questions are scaled 0-3 with 0 representing higher anxiety to 3 representing no anxiety. The depression questions are scaled from 0 indicating no depression to 3 indicating more signs of depression.
Patient reported outcomes: Hospital Anxiety and Depression Scale (HADS) | 34 Weeks
  The HADS contains 14 items that measure the frequency of anxiety and depressive symptoms over the past week. The anxiety questions are scaled 0-3 with 0 representing higher anxiety to 3 representing no anxiety. The depression questions are scaled from 0 indicating no depression to 3 indicating more signs of depression.
Patient reported outcomes: Modified Fatigue Impact Scale (MFIS) | Baseline
  The MFIS is a 21-item measure of physical, cognitive, and psychosocial impact of fatigue on daily life over the past 4 weeks. The scale ranges from 0 to 4 with 0 being never have issues regarding fatigue to 4 representing fatigue greatly affecting the participants life.
Patient reported outcomes: Modified Fatigue Impact Scale (MFIS) | 17 weeks
  The MFIS is a 21-item measure of physical, cognitive, and psychosocial impact of fatigue on daily life over the past 4 weeks. The scale ranges from 0 to 4 with 0 being never have issues regarding fatigue to 4 representing fatigue greatly affecting the participants life.
Patient reported outcomes: Modified Fatigue Impact Scale (MFIS) | 34 Weeks
  The MFIS is a 21-item measure of physical, cognitive, and psychosocial impact of fatigue on daily life over the past 4 weeks. The scale ranges from 0 to 4 with 0 being never have issues regarding fatigue to 4 representing fatigue greatly affecting the participants life.
Patient reported outcomes: Fatigue Severity Scale (FSS) | Baseline
  The FSS is a 9-item unidimensional measure of fatigue and its disabling consequences over the past week in medical populations including MS. The score is from 1 to 7 with 1 representing strongly disagreeing that fatigue has an impact on them to 7 representing strongly agreeing fatigue has an impact on the participants.
Patient reported outcomes: Fatigue Severity Scale (FSS) | 17 weeks
  The FSS is a 9-item unidimensional measure of fatigue and its disabling consequences over the past week in medical populations including MS. The score is from 1 to 7 with 1 representing strongly disagreeing that fatigue has an impact on them to 7 representing strongly agreeing fatigue has an impact on the participants.
Patient reported outcomes: Fatigue Severity Scale (FSS) | 34 Weeks
  The FSS is a 9-item unidimensional measure of fatigue and its disabling consequences over the past week in medical populations including MS. The score is from 1 to 7 with 1 representing strongly disagreeing that fatigue has an impact on them to 7 representing strongly agreeing fatigue has an impact on the participants.
Patient reported outcomes: Visual Analog Fatigue Scale (VAFS) | Baseline
  The participants will be asked to rate their global fatigue on a scale of 0-10 with 0 being the worst fatigued and 10 being normal.
Patient reported outcomes: Visual Analog Fatigue Scale (VAFS) | 17 weeks
  The participants will be asked to rate their global fatigue on a scale of 0-10 with 0 being the worst fatigued and 10 being normal.
Patient reported outcomes: Visual Analog Fatigue Scale (VAFS) | 34 Weeks
  The participants will be asked to rate their global fatigue on a scale of 0-10 with 0 being the worst fatigued and 10 being normal.
Patient reported outcomes: Short-form McGill Pain Questionnaire Revised (SF-MPQ-2) | Baseline
  The SF-MPQ has a 15-item adjective checklist that captures sensory and affective dimensions of pain experienced over the past week. Questions are scored from 0-10. Zero representing no pain and 10 representing the highest pain level.
Patient reported outcomes: Short-form McGill Pain Questionnaire Revised (SF-MPQ-2) | 17 weeks
  The SF-MPQ has a 15-item adjective checklist that captures sensory and affective dimensions of pain experienced over the past week. Questions are scored from 0-10. Zero representing no pain and 10 representing the highest pain level.
Patient reported outcomes: Short-form McGill Pain Questionnaire Revised (SF-MPQ-2) | 34 Weeks
  The SF-MPQ has a 15-item adjective checklist that captures sensory and affective dimensions of pain experienced over the past week. Questions are scored from 0-10. Zero representing no pain and 10 representing the highest pain level.
Patient reported outcomes: Pittsburg Sleep Quality Index (PSQI) | Baseline
  The questionnaire has fill in the blank questions along with questions that are rated on a scale. The scale rating is "not during the past month" to "three or more times per week."
Patient reported outcomes: Pittsburg Sleep Quality Index (PSQI) | 17 weeks
  The questionnaire has fill in the blank questions along with questions that are rated on a scale. The scale rating is "not during the past month" to "three or more times per week."
Patient reported outcomes: Pittsburg Sleep Quality Index (PSQI) | 34 Weeks
  The questionnaire has fill in the blank questions along with questions that are rated on a scale. The scale rating is "not during the past month" to "three or more times per week."

OTHER OUTCOMES:
Blood work: glucose | Baseline
  The following serum chemistry will be performed: glucose
Blood work: glucose | 17 weeks
  The following serum chemistry will be performed: glucose
Blood work: glucose | 34 Weeks
  The following serum chemistry will be performed: glucose
Blood work: insulin | Baseline
  The following serum chemistry will be performed: insulin
Blood work: insulin | 17 weeks
  The following serum chemistry will be performed: insulin
Blood work: insulin | 34 Weeks
  The following serum chemistry will be performed: insulin
Blood work: lipids | Baseline
  The following serum chemistry will be performed: lipids
Blood work: lipids | 17 weeks
  The following serum chemistry will be performed: lipids
Blood work: lipids | 34 Weeks
  The following serum chemistry will be performed: lipids
Blood work: TNF-a | Baseline
  The following serum chemistry will be performed: TNF-a
Blood work: TNF-a | 17 weeks
  The following serum chemistry will be performed: TNF-a
Blood work: TNF-a | 34 Weeks
  The following serum chemistry will be performed: TNF-a
Blood work: IL-6 | Baseline
  The following serum chemistry will be performed: IL-6
Blood work: IL-6 | 17 weeks
  The following serum chemistry will be performed: IL-6
Blood work: IL-6 | 34 Weeks
  The following serum chemistry will be performed: IL-6
Blood work: IL-17 | Baseline
  The following serum chemistry will be performed: IL-17
Blood work: IL-17 | 17 weeks
  The following serum chemistry will be performed: IL-17
Blood work: IL-17 | 34 Weeks
  The following serum chemistry will be performed: IL-17
Blood work: adiponectin | Baseline
  The following serum chemistry will be performed: adiponectin
Blood work: adiponectin | 17 weeks
  The following serum chemistry will be performed: adiponectin
Blood work: adiponectin | 34 Weeks
  The following serum chemistry will be performed: adiponectin
Blood work: leptin | Baseline
  The following serum chemistry will be performed: leptin
Blood work: leptin | 17 weeks
  The following serum chemistry will be performed: leptin
Blood work: leptin | 34 Weeks
  The following serum chemistry will be performed: leptin
Blood work: T17 | Baseline
  The following serum chemistry will be performed: T17
Blood work: T17 | 17 weeks
  The following serum chemistry will be performed: T17
Blood work: T17 | 34 Weeks
  The following serum chemistry will be performed: T17
Blood work: NFL | Baseline
  The following serum chemistry will be performed: NFL
Blood work: NFL | 17 weeks
  The following serum chemistry will be performed: NFL
Blood work: NFL | 34 Weeks
  The following serum chemistry will be performed: NFL
Blood Pressure | Baseline
  Systolic and diastolic blood pressure will be measured.
Blood Pressure | 17 weeks
  Systolic and diastolic blood pressure will be measured.
Blood Pressure | 34 Weeks
  Systolic and diastolic blood pressure will be measured.
Anthropometric Measures: Weight | Baseline
  Weight will be measured using kilograms.
Anthropometric Measures: Weight | 17 weeks
  Weight will be measured using kilograms.
Anthropometric Measures: Weight | 34 Weeks
  Weight will be measured using kilograms.
Anthropometric Measures: Height | Baseline
  Height will be measured using meters.
Anthropometric Measures: Height | 17 weeks
  Height will be measured using meters.
Anthropometric Measures: Height | 34 weeks
  Height will be measured using meters.
Anthropometric Measures: Waist circumference | Baseline
  Waist circumference will be measured using inches.
Anthropometric Measures: Waist circumference | 17 weeks
  Waist circumference will be measured using inches.
Anthropometric Measures: Waist circumference | 34 Weeks
  Waist circumference will be measured using inches.
Total Body Composition | Baseline
  Dual energy x-ray absorptiometry (DXA) Total and regional body composition will be measured on a Lunar Prodigy with enCORE software version 13.6 (GE Healthcare, Chicago, IL). Participants will undergo a total body scan requiring about 20 minutes, while lying on their back on a padded table with metal objects removed. The scan provides estimates of soft tissue attenuation ratios, fat and lean tissue mass, and bone mineral density. Individuals who are too large to scan in a single scan will be scanned twice (one scan for the left half of body, one for the right). The software is able to merge the two scans to assess total body composition. All women of child-bearing age will be required to complete a pregnancy test in the lab prior to DXA scan.
Total Body Composition | 17 weeks
  Dual energy x-ray absorptiometry (DXA) Total and regional body composition will be measured on a Lunar Prodigy with enCORE software version 13.6 (GE Healthcare, Chicago, IL). Participants will undergo a total body scan requiring about 20 minutes, while lying on their back on a padded table with metal objects removed. The scan provides estimates of soft tissue attenuation ratios, fat and lean tissue mass, and bone mineral density. Individuals who are too large to scan in a single scan will be scanned twice (one scan for the left half of body, one for the right). The software is able to merge the two scans to assess total body composition. All women of child-bearing age will be required to complete a pregnancy test in the lab prior to DXA scan.
Total Body Composition | 34 Weeks
  Dual energy x-ray absorptiometry (DXA) Total and regional body composition will be measured on a Lunar Prodigy with enCORE software version 13.6 (GE Healthcare, Chicago, IL). Participants will undergo a total body scan requiring about 20 minutes, while lying on their back on a padded table with metal objects removed. The scan provides estimates of soft tissue attenuation ratios, fat and lean tissue mass, and bone mineral density. Individuals who are too large to scan in a single scan will be scanned twice (one scan for the left half of body, one for the right). The software is able to merge the two scans to assess total body composition. All women of child-bearing age will be required to complete a pregnancy test in the lab prior to DXA scan.
Detailed body composition | Baseline
  The investigators will perform MRI to assess adipose distribution in the abdomen and thigh
Detailed body composition | 34 Weeks
  The investigators will perform MRI to assess adipose distribution in the abdomen and thigh
Neuroinflammation | Baseline
  The investigators will perform diffusion basis spectrum imaging (DBSI) MRI to assess neuroinflammation at WUSTL only
Neuroinflammation | 34 Weeks
  The investigators will perform DBSI MRI to assess neuroinflammation at WUSTL only

CONTACTS AND LOCATIONS:
Overall Officials: Brooks Wingo, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (2):
- United States (2):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Washington University, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin K, Cofield SS, Cross AH, Goss AM, Raji CA, Rinker JR, Wu GF, Blair J, Fuchs A, Ghezzi L, Green K, Pace F, Pastori G, Taylor MG, Piccio L, Wingo BC. Functional outcomes of diets in multiple sclerosis (FOOD for MS): Protocol for a parallel arm randomized feeding trial for low glycemic load and calorie restriction. Contemp Clin Trials. 2024 Aug;143:107584. doi: 10.1016/j.cct.2024.107584. Epub 2024 May 29. PMID 38821260